CLINICAL TRIAL: NCT00741637
Title: A Randomized, Placebo-Controlled Trial to Evaluate the Safety and Immunogenicity of a Single Dose Regimen of Live Attenuated Oral Cholera Vaccine (Choleragarde®) in HIV-Seropositive Adults in Thailand
Brief Title: Safety and Immunogenicity of Single Dose Choleragarde® in HIV-Seropositive Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: International Vaccine Institute (Other)
Collaborators: Vaccine Technologies Inc. (Industry); Siriraj Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CH-PR-02
Record Dates: First submitted 2008-08-25; First posted 2008-08-26 (Estimated); Last update posted 2012-03-30 (Estimated); Status verified 2012-03

CONDITIONS: Cholera; Vibrio Infections; Diarrhea
Keywords: Vibrio Cholerae; Diarrhea; Live oral Vaccines; Immunogenicity; Safety; HIV
MeSH Terms: conditions — Cholera; Vibrio Infections; Diarrhea | interventions — Peru 15

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vaccine (Experimental): Live attenuated oral CholeraGarde® (5x107 to 1x109 CFU) vaccine
  Interventions: Biological: CholeraGarde®
- Placebo (Placebo Comparator): A buffer solution containing 2.5 g sodium bicarbonate, and 1.65 g ascorbic acid.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: CholeraGarde® — Live attenuated oral Cholera vaccine
  Each vial of CholeraGarde® contains 5x107 to 1x109 CFU of Peru-15, 6.75 mg KH2PO4, and 300 mg trehalose as a lyophilized cake in 5 mL single-dose vials
  Arms: Vaccine
Biological: Placebo — A buffer solution containing 2.5 g sodium bicarbonate, and 1.65 g ascorbic acid.
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety and immunogenicity of Peru-15 (CholeraGarde®) vaccine in HIV seropositive adult population of Bangkok Thailand

DETAILED DESCRIPTION:
Cholera re-emerged in 2006 as a global threat with a 79% increase in 2006 compared to the previous year. The re-emergence of cholera increased with increasing numbers of displaced populations living in unsanitary conditions. About 99% of the reported cases were from Africa with most of the deaths reported also from this region. Case fatality rate has increased worldwide to 2.7% however, certain areas in Africa reported as much as 30% case fatality [WER 2007]. These figures are believed to be underestimates and that as many as 120 000 deaths due to cholera are estimated to occur each year [WER 2001]. Underreporting is common due to inconsistencies in the definition of cholera and limitations of surveillance, however some countries do not report due to fear of international sanctions. In 2007, the International Health Regulation came into effect wherein trade and economic sanctions should no longer be imposed in countries reporting cholera but rather encourage open reporting so as to contain and prevent the spread of cholera epidemics [WER 2007].

Provision of safe water and food, establishment of adequate sanitation, and implementation of personal and community hygiene constitute the main public health interventions against cholera. These measures cannot be fully implemented in the near future in most cholera-endemic areas. A safe, effective, and affordable vaccine would be a useful tool for cholera prevention and control.

Considerable progress has been made during the last decade in the development of new generation oral vaccines against cholera. These have already been licensed in some countries and are now being considered for wider public health application. The World Health Organization recently recommended that the newer generation cholera vaccines be considered in certain endemic and epidemic situations, but indicated that demonstration projects are needed to provide more information about the costs, feasibility, and impact of using these vaccines [WHO Meeting 2002].

A killed oral cholera vaccine (Dukoral™) has long been available internationally, however its 2-dose schedule, the use of a buffer and the cost of the vaccine have long impeded its use in public health settings. A live oral vaccine (Orochol™), although internationally licensed is currently not available in the market. This vaccine is only available for use in children older than 6 years old and adults. Despite the immunogenicity and efficacy in challenge studies in North American volunteers [Tacket CO 1999], in a field trial of this vaccine in an endemic area in Indonesia, no protective efficacy was detected during the period of observation [Richie EE 1994].

A need exists for an improved cholera vaccine that is more thermostable and may be used in endemic countries in younger age groups. This new generation live oral cholera vaccine must be administered in a single-dose regimen, be thermostable, confer high grade long-term protection and may be given to children below 2 years of age through mass immunization campaigns or through the EPI. In the Diseases of the Most Impoverished Programme (DOMI) of the IVI, Peru-15 (CholeraGarde®) was identified as the most promising of all the vaccine candidates. It is a live oral attenuated cholera vaccine derived from V. cholerae O1 El Tor Inaba strain that was first isolated in Peru in 1991 [Taylor DN 1994]. This has the advantage of having the same biotype as the current pandemic strain. Peru-15 has been attenuated by several genetic modifications and deletions. By the deletion of the ctx A and the rtxA genes, it has been rendered unable to encode for cholera toxin subunit A and RTX toxin making it non-toxigenic; by the inactivation of the recA gene and deletion of the attRS1 sequences, it has been made unable to integrate exogenous DNA making it non-recombination and by the absence of the potentially inflammatory flagella it has been rendered non-motile [Taylor DN 1994, Kenner 1995]. Phase I and II studies have been performed in North American volunteers where it was found to be safe and immunogenic [Kenner 1995, Sack 1997] . Furthermore, the vaccine strain isolated from the stools of volunteers retained its non-motile characteristic. In a challenge study among North American volunteers, Peru-15 provided 100% protection against moderate and severe diarrhoea, and 93% against any diarrhoea [Cohen 2002].

This vaccine underwent phase I and II studies in a cholera-endemic area in Matlab, Bangladesh in three age groups: adults aged 18 - 45 years, children aged 2 - 5 years and infants aged 9 - 23 months [Qadri 2007]. In these studies, the vaccine has been shown to be safe and elicit vibriocidal responses among all age groups. Only 1 of 20 adults and 8 of 140 children vaccine recipients excreted the vaccine strain. Analysis of the strains isolated revealed that the strains remained unchanged in phenotypic and genotypic properties after passage in the stool.

Although this vaccine can be given as a single dose, and appears to be immunogenic in infants, the vaccine requires stringent cold storage conditions at -20ºC. Avant Immunotherapeutics Inc., manufacturers of Peru-15, is currently reformulating the vaccine in order to make it more thermostable. In order to assess whether this vaccine is as safe and immunogenic as the previous formulation, this lyophilized formulation will need to undergo clinical testing in an endemic community.

The International Vaccine Institute (IVI) through the Cholera Vaccine Initiative (CHOVI) together with Avant Immunotherapeutics Inc., manufacturers of the Peru-15 vaccine, have negotiated an agreement that allows clinical trials to be performed in cholera-endemic countries, including, India, Bangladesh, and Thailand. This will eventually enable licensure and facilitate the international use of this vaccine by obtaining a WHO recommendation for its global use. This single dose vaccine may easily be used in endemic countries and deployed at times when outbreaks are likely to occur.

Because cholera tends to occur in areas where the seroprevalence of HIV is also high, safety and immunogenicity of any vaccine against cholera must be established among HIV infected individuals. There is limited data regarding the use of oral cholera vaccines among HIV seropositive individuals. A study in Beira, Mozambique, an area with a 20-30% HIV seroprevalence revealed that the killed oral rBS-WC vaccine may be effective against cholera [12]. However, specific data on HIV status and safety of the vaccine was not determined in the study. The live attenuated CVD 103 HgR vaccine was found to be equally safe among HIV seropositive and HIV seronegative individuals in Mali. The vaccine however was found to result in attenuated immune response among HIV seropositive individuals [Perry 1998].

In order for the Peru-15 cholera vaccine to be used extensively in cholera outbreaks or in cholera endemic settings where HIV co-exists, safety and immunogenicity must first be established among HIV-seropositive individuals.

To gain approval for use in the developing world, a single-dose of CholeraGarde® will have to confer high levels of protective efficacy for three years when given to endemic populations 9 months and older. However, before undertaking a phase III efficacy trial, a series of phase II clinical studies need be conducted in order to confirm safety and immunogenicity of the vaccine. Since cholera and HIV co-exist in some areas of the world, safety and immunogenicity of the Peru-15 vaccine must be established among HIV seropositive individuals.

ELIGIBILITY:
Inclusion Criteria:

HIV-seropositive, non-pregnant adults, aged 18 - 45 years old who have been on standard highly active antiretroviral therapy (HAART) for at least 6 months prior to enrollment or who have never started HAART regimen will be recruited in the study.

All subjects must satisfy the following criteria at study entry:

1. Male and female HIV seropositive adults aged 18 to 45 years old who have given the written informed consent.
2. Will comply with the requirements of the protocol (i.e. available for follow-up visits and specimen collection).
3. CD4 T-lymphocyte count >500/mm3 for at least 6 months prior to inclusion

Subjects that have never started HAART regimen must satisfy the following additional criteria at study entry.

1. Asymptomatic HIV infection as determined by: Medical history, Physical examination, Laboratory tests, Clinical judgment of the investigator

Subjects that have been on standard highly active antiretroviral therapy (HAART) for at least 6 months prior to enrollment must satisfy the following additional criteria at study entry.

1. History of CD4 nadir >150/mm3
2. Viral load (HIV-1 RNA levels) <200 copies/mL for at least 6 months prior to inclusion

Exclusion Criteria:

The following criteria should be checked at the time of study entry, if any of the following is present then the subject will be excluded from the study:

1. Overt signs of immunodeficiency e.g. oral thrush, rapid weight loss, recurrent pneumonia (i.e. Stage 3 or 4 of the WHO clinical staging system for HIV infection and disease in adults and adolescents
2. Ongoing serious chronic illness (e.g. with signs of cardiac or renal failure)
3. Abdominal pain or cramps, loss of appetite, nausea, general ill-feeling or vomiting in the past 24 hours
4. Presence of V. cholerae 01 or 0139, Shigella, or Cryptosporidium in stool at baseline
5. Intake of any anti-diarrhoeal medicine in the past week
6. Acute disease one week prior to enrollment, with or without fever. Temperature ≥38ºC (oral or otic) warrants deferral of the vaccination pending recovery of the subject
7. Receipt of antibiotics in the past 2 weeks
8. Receipt of live or killed enteric vaccine in the last 4 weeks
9. Receipt of killed oral cholera vaccine in the past
10. Diarrhea (3 or more loose stools within a 24-hour period) 6 weeks prior to enrollment
11. One or more episodes of diarrhea lasting for more than 2 weeks in the past 6 months
12. One or more episodes of abdominal pain lasting for more than 2 weeks in the past 6 months
13. Receipt of blood, blood products or a parenteral immunoglobulin preparation in the previous 6 months
14. Receipt of any immunosuppressive therapy during the past 6 months
15. A woman pregnant or planning to become pregnant during the period of subject's participation
16. Any condition which in the opinion of the investigator, might interfere with the evaluation of the study objectives

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2010-07; Primary Completion 2011-04 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects receiving CholeraGarde® or placebo with any of the following events within 7 days of dosing: Gas, headache, vomiting, abdominal cramps, myalgias, diarrhea, fever | 0,1,2,3,4,5,6,7,14,30,90 days post intervention

SECONDARY OUTCOMES:
Proportion of subjects exhibiting 4-fold or greater rises in titers of serum vibriocidal antibodies to 01 serogroup El Tor Inaba organisms, relative to baseline, one week after a single dose of CholeraGarde® or placebo | 0,1,2,3,4,5,6,7,14,30,90 days post vaccination
Proportion of subjects given CholeraGarde® or placebo with any of the following adverse events | 30 minutes after adminstration and throughout the trial
Geometric mean serum vibriocidal IgG antibody titers measured at baseline and one week after a single dose of CholeraGarde® or placebo | One week
Proportion of subjects given CholeraGarde® or placebo with fecal excretion of CholeraGarde® | At 3, 7, 14, and 30 days post-dosing
Mean HIV viral load (copies/ml) increases, with CholeraGarde® or placebo | relative to baseline, at 7, 30, and 90 days post-dosing
Mean CD4 lymphocyte count, with CholeraGarde® or placebo | relative to baseline, at 90 days post-dosing

CONTACTS AND LOCATIONS:
Overall Officials: Winai Ratanasuwan, MD, MPH, Principal Investigator — Siriraj Hospital
Locations (1):
- Department of Preventive and Social Medicine Siriraj Hospital, Bangkok, Thailand